CLINICAL TRIAL: NCT05881356
Title: Understanding the Patient Perspective: An Observational Study on Experiences of OCD Clinical Trial Patients
Brief Title: Discovering Factors in the Clinical Study Journey of Patients With OCD
Status: Recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 91191727
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: OCD; Obsessive-Compulsive Disorder
Keywords: OCD; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research aims to collect comprehensive data on the clinical trial experience of OCD patients. Its goal is to identify the factors that limit patients' ability to join or complete a trial successfully. Clinical trial participation often favors specific demographic groups, and limited research exists on the impact of trial attributes on participation. Therefore, this study aims to analyze data from various demographic groups and identify any recurring trends that could provide valuable insights for future OCD patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Participant has a diagnosis of OCD.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

Exclusion Criteria:

* Pregnant or lactating woman
* Enrolled in another research study
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with OCD who are actively considering involvement in an observational clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of participants who decide to enroll in a OCD clinical study. | 3 months
Number of OCD patients who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hirschtritt ME, Bloch MH, Mathews CA. Obsessive-Compulsive Disorder: Advances in Diagnosis and Treatment. JAMA. 2017 Apr 4;317(13):1358-1367. doi: 10.1001/jama.2017.2200. PMID 28384832
- [Background] Albert U, Marazziti D, Di Salvo G, Solia F, Rosso G, Maina G. A Systematic Review of Evidence-based Treatment Strategies for Obsessive- compulsive Disorder Resistant to first-line Pharmacotherapy. Curr Med Chem. 2018;25(41):5647-5661. doi: 10.2174/0929867325666171222163645. PMID 29278206
- [Background] Bidlack JM, Lockshin RA. Evolution of LDH isozymes during programmed cell death. Comp Biochem Physiol B. 1976;55(2):161-6. doi: 10.1016/0305-0491(76)90223-6. No abstract available. PMID 963971

DOCUMENTS (1):
  • Informed Consent Form (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT05881356/ICF_000.pdf